CLINICAL TRIAL: NCT04824430
Title: Assessment of Uterine Access, Uterine Patency and Intrauterine Adhesions (IUA) 3, 6 and 12 Months Following Endometrial Ablation: A Prospective Single-Center Observational Study
Brief Title: Assessment of Uterine Access, Uterine Patency and Intrauterine Adhesions Following Endometrial Ablation
Status: Completed | Type: Observational
Sponsor: Rejoni Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: EA 21-001
Record Dates: First submitted 2021-03-24; First posted 2021-04-01 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Intrauterine Adhesion
MeSH Terms: conditions — Gynatresia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- SLH 3M: Second look hysteroscopy (SLH) performed 3 months post-ablation
- SLH 6M: Second look hysteroscopy (SLH) performed 6 months post-ablation
- SLH 12M: Second look hysteroscopy (SLH) performed 12 months post-ablation

SUMMARY:
The objective of this study is to gain information concerning the acute and longer-term morphological changes within the uterus following endometrial ablation. Hysteroscopic evaluation of the uterine cavity will be used to determine if physical access and the ability to systematically assess the post-ablation uterine cavity were preserved. The presence, location and severity of intrauterine adhesions will be documented in participants who are 3, 6 and 12 months from their standard of care endometrial ablation.

DETAILED DESCRIPTION:
Prospective single center observational study. Up to 30 subjects will be enrolled (up to 10 subjects per time point). Patients who sign the Institutional Review Board (IRB) approved consent form who have undergone endometrial ablation within the prior 14 months from time of consent will be asked to participate in this study. Patients meeting all eligibility criteria will undergo either a 3, 6 or 12 month diagnostic second look hysteroscopy (SLH) as assigned by the Investigator depending on the duration of time between the ablation and the signature date of the informed consent (up to 10 subjects for each time point). A diagnostic SLH will be performed for scoring of intrauterine adhesions by the investigator and an independent reviewer. The ability to access the uterine cavity (or not) will be documented.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal female patients ≥ 18 years of age
* Patient has undergone endometrial ablation within the prior 14 months.
* There were no contraindications for endometrial ablation as specified in Ablation System labeling
* Patient agrees to undergo an SLH either at 3, 6 or 12 months post-ablation
* Patient abstained from any form of hormonal contraception including an IUD after the ablation and through the period that the SLH is performed.
* Patient has signed the IRB approved informed consent.

Exclusion Criteria:

* Additional intrauterine procedures performed between time of endometrial ablation and the SLH; e.g., endometrial and/or myometrial resection.
* IUD in situ
* Pregnant (positive urine pregnancy test) or lactating
* Active sexually transmitted infection or genital infection, or other clinically significant active and/or systemic infection per clinical or laboratory examinations at the time of endometrial ablation procedure or second look hysteroscopy (e.g., cervicitis, vaginitis, endometritis, or salpingitis).
* Systemic steroid within 1 week of endometrial ablation
* Previous adhesiolysis procedure or diagnosis of Asherman's disease.
* No noted clinically significant uterine anomalies at the time of the ablation (e.g., septate uterus or other anomalies that distorts the uterine cavity)
* Any other condition that in the opinion of the investigator could represent an increased risk for the subject, affect the primary outcomes of this study and/or impact the subject's ability to comply with protocol requirements.
* Participating or considering participation in a clinical trial of another investigational drug or device during this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women who meet eligibility criteria having undergone a prior endometrial ablation 3, 6 or 12 months prior to the second look hysteroscopy
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2021-07-22 (Actual); Study Completion 2021-07-22 (Actual)

PRIMARY OUTCOMES:
Incidence of Intrauterine Adhesions (IUA) | 3, 6 or 12 months post-ablation

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Basinski, MD, Principal Investigator — Basinski and Juran MDs
Locations (1):
- Basinksi and Juran, MD's, Newburgh, Indiana, United States

IPD SHARING:
Plan to Share IPD: No